CLINICAL TRIAL: NCT01309542
Title: A 10 Month Open-Label Evaluation Of The Long-Term Safety Of DVS-233 SR In Outpatients With Major Depressive Disorder.
Brief Title: Long-Term Safety Of DVS-233 SR In Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3151A1-303; B2061069
Record Dates: First submitted 2011-02-24; First posted 2011-03-07 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; desvenlafaxine; antidepressant
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DVS (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate

INTERVENTIONS:
Drug: Desvenlafaxine Succinate — Tablet were taken at a daily dose of 200 to 400 mg/day for a duration up to 10 months
  Other Names: DVS-233 SR

SUMMARY:
The study evaluated the long-term safety of Desvenlafaxine Succinate (DVS) Slow Release (SR) during open-label treatment in adult outpatients who had a primary diagnosis of major depressive disorder (MDD). The study also evaluated the long-term response of subjects receiving DVS SR for clinical global evaluation, functionality, general well-being, pain, and absence of depressive symptoms (remission).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who have completed double-blind therapy in a phase 3 DVS-233 SR short-term study for the indication of MDD, including scheduled evaluations, with no major protocol violations and no study events that, in the opinion of the investigator, would preclude the subject's entry into the long-term, open-label study.
* Sexually active individuals participating in the study must use a medically acceptable form of contraception during the trial and for at least 15 days after the last dose of study drug.

Exclusion Criteria:

* Clinically important abnormalities on baseline physical examination, or any unresolved clinically significant abnormalities on ECG, laboratory test results, or vital signs recorded in a previous phase 3 DVS-233 SR short-term study for the indication of MDD. Any exception must be discussed with and granted by the sponsor.
* Significant risk of suicide based on clinical judgment, including common suicidal thoughts, and suicide being considered as a possible solution, even without specific plans or intention.
* Presence of clinically important hepatic or renal disease or other medical disease that might compromise the study or be detrimental to the subject (eg, clinically important cardiac arrhythmia, uncontrolled diabetes, uncontrolled hypertension, seizure disorder, myocardial infarction, neurologic disorder, acute illness, neoplastic disorder).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1403 (Actual)
Dates: Start 2003-08; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Number (%) of Subjects Reporting Adverse Events during Treatment | 10 months
Number (%) of Subjects With Changes in Vital Signs (Blood Pressure, Pulse Rate, Weight) of Potential Clinical Importance | 10 months
Number (%) of Subjects With Laboratory Test Results (Hematology, Blood Chemistry, Lipid Profile, Urinalysis) of Potential Clinical Importance | 10 months
Number (%) of Subjects With Electrocardiogram Results (Heart Rate, QTc interval) of Potential Clinical Importance | 10 months

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating scale - 17 items version - (HAM-D17) mean score from baseline | 10 months
Change in Montgomery Asberg Depression Rating Scale (MADRS)mean score from baseline | 10 months
Change in Clinical Global Improvement Scale-Severity (CGI-S)mean score from baseline | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (117):
- United States (53):
  - Birmingham Research Group Inc., Birmingham, Alabama
  - Pivotal Research Centers 13128 North 94th Drive, Suite 200, Mesa, Arizona
  - Pivotal Research, Peoria, Arizona
  - Southwestern Research, Inc., Beverly Hills, California
  - Feighner Research Institute, Chula Vista, California
  - California Clinical Trials Medical Group, Inc., Glendale, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pacific Clinical Research, Orange, California
  - UCSD Department of Psychiatry Psychopharmacology Research, San Diego, California
  - Southwestern Research, Inc., Tustin, California
  - Alpine Clinical Research Center, Inc., Boulder, Colorado
  - Feiger Health Research Center, Lakewood, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - New Britain General Hospital, New Britain, Connecticut
  - The George Washington University Medical Center, Washington D.C., District of Columbia
  - CORE Research, Inc.1006 NW 14, Leesburg, Florida
  - Lifestream Behavioral Center, Leesburg, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Miami Research Associates, Inc., South Miami, Florida
  - Comprehensive NeuroScience, Inc., St. Petersburg, Florida
  - Kolin Research Group 1065 West Morse Blvd. Suite 202, Winter Park, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Atlanta Institute of Medicine & Research, Marietta, Georgia
  - Carman Research, Smyrna, Georgia
  - Radiant Research - Chicago, Chicago, Illinois
  - Ingenium Clinical Research, Libertyville, Illinois
  - Capital Clinical Research Associates, LLP, Rockville, Maryland
  - DuPont Clinical Research, Inc., Rockville, Maryland
  - Institute for Health Studies, Okemos, Michigan
  - Creighton University, Omaha, Nebraska
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - CRI Worldwide, LLC, Clementon, New Jersey
  - Social Psychiatry Research Institute, New York, New York
  - The Medical Research Network, New York, New York
  - Anxiety & Depression Clinic, The Bronx, New York
  - Piedmont Neuropsychiatry, Charlotte, North Carolina
  - Hartford Research Group, Cincinnati, Ohio
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Southeastern Pennsylvania Medical Institute, Havertown, Pennsylvania
  - RI Mood & Memory Research Institute, East Providence, Rhode Island
  - Southeast Health Consultants, LLC, Charleston, South Carolina
  - Carolina Clinical Research Services, Columbia, South Carolina
  - FutureSearch Trials, Austin, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Research Testing, Inc., Houston, Texas
  - Radiant Research Salt Lake City, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington
  - Center for Anxiety and Depression, Seattle, Washington
  - Northbrooke Research Center, Brown Deer, Wisconsin
- Estonia (3):
  - West Tallinn Central Hospital, Tallinn, Estonia
  - Jaanson-Lääne Outpatient Clinic, Tartu, Estonia
  - Viljandi Hospital Foundation Psychiatric Clinic, Viljandi, Estonia
- Finland (12):
  - Psychiatric Research Clinic of Kupio, Kuopio, Finland
  - Psykoforum OY, Tampere, Finland
  - Psykiatripalvelu AT Oy, Espoo
  - FF Research, Helsinki
  - Mehilainen clinic, Helsinki
  - Mehiläinen, HUCH, Helsinki
  - Hakaniemen Lääkäriasema, Helsinki
  - Satakunnanpsykiatripalvelu, Rauma
  - MediRoi Oy, Rovaniemi
  - Psychiatric Research clinic of Salo, Salo
  - Länsi-Suomen Erikoislaakaripalvelu Oy, Turku
  - Turku Psychiatric Services Aurakatu 14 B 3 Krs, Turku
- France (12):
  - 57 rue Gamard, Joué-Les-Tours, France
  - 1, avenue du 6 Juin, Caen
  - 88 Rue Emmanuel Liais, Cherbourg
  - Centre Médico-Psychologique, Dole
  - Résidence St Michel, Douai
  - Immeuble Impérial, La Valette-du-Var
  - 16 avenue Robert Schuman, Mulhouse
  - 3 rue Marceau, Nantes
  - Office of Dr Marce Zins-Ritter, Orvault
  - 22 rue de Nemours, Rennes
  - 7, rue Georges Politzer, Saint-Cyr-l'École
  - 13 place Gaston Paillhou, Tours
- Germany (6):
  - emovis GmbH, Berlin
  - Praxis fuer Psychiatrie, Dr. Franz, Berlin
  - Praxis für Psychiatrie, Dr. Alexander Schulze, Berlin
  - Psychiatrische Praxis Dr. Hans-Peter Wunderlich, Dresden
  - Praxis f. Neurologie u. Psychiatrie Dr. Lutz D. Lohse, Dresden
  - Dr. D. Backhaus, Hildesheim, Hildesheim
- Latvia (3):
  - Psychoneurological hospital of Jelgava, Dept No12, Jelgava, Latvia
  - Riga Mental Health Care Center, Dept of Psychiatry, Riga, Latvia
  - Strenci Psychiatric Hospital, Strenči, Latvia
- Lithuania (3):
  - Medical center Neuromeda, Kaunas, Lithuania
  - Klaipeda Psychiatry Hospital, Klaipėda, Lithuania
  - Vilnius Mental Health Care, Vilnius, Lithuania
- Poland (11):
  - SP ZOZ Swietokrzyskie Centrum Psychiatrii w Morawicy, Gmina Morawica, Poland
  - Poradnia Zdrowia Psychicznego w Chelmnie, Chełmno
  - Akademii Medycznej w Bialymstoku, Choroszcz
  - Wojewodzki Szpital Psychiatryczny, Gdansk
  - Poradnia Zdrowia Psychicznego, Kutno
  - Specjalistyczny Psychiatryczny ZOZ w Lodzi, Lodz
  - Wojewodzki Szpital dla Nerwowo i Psychicznie Chorych, Lubiąż
  - Wojewodzki Osrodek Lecznictwa Psychiatrycznego w Toruniu, Torun
  - Wojewodzki Osrodek Lecznictwa Psychiatrycznego, Torun
  - Inventiva Biomedical and Sport Research Sp. z o.o., Tuszyn
  - NZOZ Centrum Zdrowia Psychicznego, Wroclaw
- Serbia and Montenegro (2):
  - Klinicko-bolnicki centar Dr Dragisa Misovic - Dedinje, Belgrade
  - Institut za mentalno zdravlje, Beograd
- Slovakia (3):
  - University Hospital Bratislava, Bratislava
  - Nemocnica s poliklinikou Liptovsky Mikulas, Liptovský Mikuláš
  - General Hospital in Trencín, Trenčín
- South Africa (9):
  - Westville Hospital, Westville, Durban
  - Vista Clinic, Pretoria, Gauteng
  - Westdene Research Centre, Bloemfontein, Republic of South Africa
  - Vista Clinic, Pretoria, Republic of South Africa
  - Dey Clinic, Pretoria, Republic of South Africa
  - Paarl Medical Centre, Paarl, Western Cape
  - Knighton Surgery, Cape Town
  - 2B Tre Mondi Office Park, Somerset West
  - Welkom Mediclinic, Welkom

REFERENCES:
- [Derived] Tourian KA, Pitrosky B, Padmanabhan SK, Rosas GR. A 10-month, open-label evaluation of desvenlafaxine in outpatients with major depressive disorder. Prim Care Companion CNS Disord. 2011;13(2):PCC.10m00977. doi: 10.4088/PCC.10m00977blu. PMID 21977353
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-303&StudyName=Long-Term%20Safety%20Of%20DVS-233%20SR%20In%20Patients%20With%20Major%20Depressive%20Disorder